CLINICAL TRIAL: NCT02456987
Title: The Feasibility, Usability, Acceptability, and Clinical Utility of a Virtual Reality Intervention in the Inpatient Setting
Brief Title: Virtual Reality in Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Brennan Spiegel, Director, Health Services Research, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00039751
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients that qualify for the intervention will receive the Samsung Gear virtual reality experiences and will participate in a brief survey about their opinions and preferences once the experiences are completed.
  Interventions: Device: Samsung Gear
- Control (No Intervention): Age and sex matched control participants will be asked to answer a series of satisfaction questions after the study recruitment period is over. These individuals will have been inpatients during the same time as the intervention participants.

INTERVENTIONS:
Device: Samsung Gear — Intervention arm will be exposed to a series of virtual reality experiences using the Samsung Gear hardware one time during their inpatient stay at Cedars-Sinai.
  Arms: Intervention

SUMMARY:
This study is being conducted as a pilot to test the feasibility, usability, acceptability, and clinical utility of using a virtual reality (VR) immersion experience in the inpatient setting. In addition to determining whether the patients enjoy the experience and would like to participate in a future more tailored immersion in virtual reality, we will be attempting to determine whether there are any positive impacts on their visit, including a distraction from their pain or anxiety associated with their procedures or the reason they have been admitted to the hospital.

Because the inpatient population at Cedars-Sinai Medical Center (CSMC) is dynamic and diagnostically diverse, we intend to develop a series of VR interventions that broadly address patient concerns. VR has only been tested in select patient populations, so we are equally interested in the feasibility of deploying VR across the inpatient hospital environment as we are in demonstrating some effectiveness in reducing pain and anxiety, and improving satisfaction.

The present study has the following aims:

1. Adapting existing VR environments for inpatients with a variety of impairments, utilizing cost-effective VR hardware (Phase 1).
2. Assess the usability and acceptability of the VR equipment and software by hospital inpatients by conducting qualitative interviews (Phase 2).
3. Assess the clinical utility of the VR intervention by measuring patient reported outcomes using a modified care satisfaction survey, administered to inpatients receiving VR and a matched control sample (Phase 3).

Concerning Aims 2 and 3, we hypothesize the following:

1. Inpatients will find the VR intervention helpful and enjoyable, and will believe that its benefits outweigh any difficulties encountered using the hardware or software.
2. Inpatients who are exposed to the VR intervention will report significantly improved pain management, greater satisfaction with their inpatient visit, and greater overall health compared to matched control inpatients that were not exposed to VR.

DETAILED DESCRIPTION:
Recent advances in Virtual Reality (VR) technology have made it possible for researchers to develop interventions for a wide variety of disease states, including obesity, pain, impaired motor functioning, and anxiety. Over the last decade, improvements in software and hardware design, as well as associated cost reductions, have made VR a practical tool for widespread use, rather than an expensive novelty. Interventions that would not be possible or practical in the real world have been developed in the virtual world, resulting in immersive multi-sensory (primarily audio-visual) experiences that can distract patients from painful experiences and motivate them to achieve personal goals.

VR environments allow patients to visualize non-disease states, and practice living more healthily, whether the focus is stroke rehabilitation, exposure therapy for social anxiety, or simply interacting with the world with reduced pain levels. A number of studies have demonstrated the efficacy of VR interventions, and all of them are built around this basic premise. For example, a meta-analysis of diagnosis-specific exposure therapies for anxiety disorders - PTSD, agoraphobia/panic disorder, social anxiety, and animal phobias) reports large effects (Cohen's Q-statistic >0.80) for VR interventions on symptom reports at therapy termination.1 Similarly, a meta-analysis of post-stroke motor rehabilitation VR interventions reports that, in observational studies, patients experience significantly reduced impairment (14.7%) and improved motor functioning (20.1%).

Hospital inpatients will most likely benefit from VR as a distraction from acute pain during procedures, painful drug infusions, adverse side effects of treatments, or from boredom and inactivity, which could lead to increased reports of distress and reduced satisfaction with care. Several areas of research may provide a useful model for bringing VR distraction interventions to all types of hospital inpatients. A recent review by Li and colleagues (2012) highlighted advances in these treatment areas.

To date, the most widely studied form of VR interventions is the reduction of pain and anxiety associated with burn care. Compared to use of analgesic medication alone, patients who use VR distraction interventions in combination with analgesic drugs have reported reduced pain and distress during burn wound care across most studies, and both lower pain ratings and increased range of motion during physical therapy in some studies. Use of a VR distraction environment called SnowWorld - developed by H.G. Hoffman and colleagues, and employed across many of these studies - allows burn patients to move through ice canyon and play with snow. Additions of VR hypnosis and relaxation modules to SnowWorld have also been tested in burn patients, with mixed results; patients undergoing hypnosis reported lower pain and anxiety levels, but those undergoing relaxation while receiving morphine reported higher pain levels.

Studies of cancer patients have demonstrated some efficacy for use of VR in patients receiving chemotherapy and lumbar punctures. Although pain scores are often reduced in a direction favoring the use of VR, studies to date have not demonstrated conclusive, long term benefits for symptom reduction. However, patients do report short perceived time in treatment, reduced physiological arousal during treatment, and lower perceived pain during treatment.

During routine medical procedures, VR delivered via a head-mounted display demonstrated some promising effects. In a study of outpatients having blood drawn, those receiving the most immersive VR reported lower levels of moderate to severe pain. In a similar study of patients having an IV placed for CT scan contrast, those receiving VR reported no change in pain level, compared to standard care patients who reported a four-fold increase in pain.

VR has also been used for the treatment of chronic pain. In a sample of adults with chronic neck pain, use of a VR mirror visual feedback environment resulted in promising but non-significant reported pain reductions. In another study of patients with chronic neck pain, a single session of VR that encouraged increased range of motion (by spraying at flies).

Notably, many of these studies (except for chronic neck pain patients) were conducted using child and adolescent populations. This group may be more receptive to VR, given common exposure to video games and screen-based entertainment. Nevertheless, the use of VR for all patients should be studied further, as the intervention may present a novel and cost-effective method of improving patient experiences and satisfaction.

VR interventions have been used as distractions or diversions during medical procedures. This study will be one of the first to test the feasibility of deploying low-cost VR interventions in a nonsurgical inpatient hospital setting. The VR hardware configuration and all software is currently being developed by AppliedVR, a leader in the development of medical applications for virtual reality technology, including interventions for weight loss and health, safety training, education, and personal development.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the goals of the study and provide informed consent
* Any Inpatient at CSMC ISP, admitted between June 2015 and 31 December 2016, who is not excluded due to criteria listed below.
* At least 18 years of age
* English speaking

Exclusion Criteria:

* Unable to consent to study due to cognitive difficulty
* Current diagnosis of epilepsy, dementia, or other neurological disease that may prevent use of VR hardware and software
* Vision requiring correction with eyeglasses (except nearsightedness, which can be accommodated by the Gear VR goggles)
* Sensitivity to flashing light or motion*
* Recent stroke
* Transplant patient
* Patient on ventilator, BiPAP, or other breathing assistance equipment
* Recent injury to the eyes, face, neck, or arms that prevents comfortable use of VR hardware or software*
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Qualitative Survey Instrument | up to 10 min (Immediately following intervention)
  Patients involved in the intervention will be asked a series of qualitative questions asking about their overall experience of the virtual reality intervention as well as the different virtual experiences and how they might change them.

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Spiegel, MD, MSHS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Derived] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654